CLINICAL TRIAL: NCT06014359
Title: Effect of Preoperative Nebulized Dexmedetomidine on Hemodynamic Changes in Morbidly Obese Patients Undergoing Laparoscopic Bariatric Surgery.
Brief Title: Preoperative Nebulized Dexmedetomidine on Hemodynamic Changes in Laparoscopic Bariatric Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdelhamed Ibrahim Abdelhamed Badreldin, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS150/4/23
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Dexmedetomidine; Hemodynamics; Laparoscopic Bariatric Surgery
MeSH Terms: interventions — Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients of this group will be Nebulized with 3 mL of 0.9% saline 15 minutes before shifting the patients to operation room with face mask 6 L/min in sitting position.
  Interventions: Drug: Saline
- Study group (Experimental): Patients of this group will be Nebulized with Dexmedetomidine (1 mcg/kg) in 3mL of 0.9% saline 15 minutes before shifting the patients to operation room with face mask 6 L/min in sitting position.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Saline — Patients will be Nebulized with 3 mL of 0.9% saline 15 minutes before shifting the patients to operation room with face mask 6 L/min in sitting position.
  Arms: Control group
Drug: Dexmedetomidine — Patients will be Nebulized with Dexmedetomidine (1 mcg/kg) in 3mL of 0.9% saline 15 minutes before shifting the patients to operation room with face mask 6 L/min in sitting position.
  Arms: Study group

SUMMARY:
This randomized study aims to evaluate the effect of preoperative dexmedetomidine nebulization on blunting hemodynamic response for laryngoscope, intubation and pneumoperitoneum in morbidly obese patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is an α -2 adrenergic agonist that has been proven to attenuate the hemodynamic response to intubation and pneumoperitoneum along with dose sparing effect on opioids and propofol .It has been used in multiple routes such as intravenous, intramuscular, oral, nasal, or intrathecal routes .Inhalation of nebulized drug is noninvasive and associated with high bioavailability .Nebulized Dexmedetomidine may offer an attractive alternative to both intravenous as well as intranasal routes of administration because drug deposition following nebulization takes place over nasal, buccal, as well as respiratory mucosa.

ELIGIBILITY:
Inclusion Criteria:

* This study will include 90 adult morbidly obese patients of both sex with BMI (40-50), (ASA) III physical status, aged between 18 -50 years scheduled for elective laparoscopic bariatric surgery under general anesthesia.

Exclusion Criteria:

1. Patient's refusal.
2. Decompensated hepatic or renal or cardiac disease.
3. Expected difficult airway management.
4. Uncontrolled hypertension.
5. Psychiatric disease.
6. Sever pulmonary disorders.
7. Patients on opioid, alcohol, beta-blockers or allergy to any of the study drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-27 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic response to laryngoscope, and pneumoperitoneum. | Intraoperative
  Heart rate (HR) and non-invasive mean arterial blood pressure (MAP) changes before nebulization, after nebulization, immediately after induction, after intubation at (1-3-6 minutes), post-pneumoperitoneum(T0) then every 15 minutes till end of the surgery.

SECONDARY OUTCOMES:
Degree of sedation | Just after nebulization
  Ramsay Sedation Scale).
  1. Awake; agitated or restless or both.
  2. Awake; cooperative, oriented, and tranquil.
  3. Awake but responds to commands only.
  4. Asleep; brisk response to light glabellar tap or loud auditory.
  5. Asleep; sluggish response to light glabellar tap or loud auditory stimulus.
  6. sleep; no response to glabellar tap or loud auditory stimulus.
Amount of opioid consumption | 24 hours postoperative
  After assessment of pain scores, when NRS measures more than (3), patients will receive 3 mg morphine, which can be repeated considering that the total daily consumption of morphine never exceeds 20 mg.
Amount of fentanyl consumption | Intraoperative
  Additional doses of fentanyl (50 mcg) will be given if HR and MAP unexplained increased more than 20% from base line during surgery, and total consumption of fentanyl will be recorded, patients in whom the first attempt of tracheal intubation have failed will be rulled out from the study.
Postoperative pain | 24 hours postoperative
  Postoperative pain will be measured using numerical rating scale (NRS) where (0 = no pain, 10 = the worst possible pain), postoperative pain will be assessed 30 minutes postoperatively then at ( 2,4,6,12,18,24 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Abdelhamed I Badreldin, MBBCH, Principal Investigator — Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt.
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author